CLINICAL TRIAL: NCT04410783
Title: The ED-SED Pilot: a Multicenter, Before-After Study to Improve Sedation in the Emergency Department
Brief Title: The Emergency Department Sedation Pilot Trial
Acronym: ED SED Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: University of Iowa (Other); Cooper University Health Care (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Brian Fuller, Associate Professor of Anesthesiology and Emergency Medicine, Washington University School of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 201909100; R34HL150404 (NIH)
Record Dates: First submitted 2020-05-20; First posted 2020-06-01 (Actual); Results first posted 2022-12-28 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Mechanical Ventilation; Respiratory Failure
Keywords: Sedation; Mechanical Ventilation; Emergency Department; RASS
MeSH Terms: conditions — Respiratory Insufficiency; Emergencies | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: This is a prospective, before-and-after study, and there will be no randomization process.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Before group (Other): Mechanically ventilated emergency department patients receiving standard post-intubation sedation prior to an educational initiative on the importance of ED-based targeted sedation
  Interventions: Other: Standard post intubation sedation practices
- After group (Other): Mechanically ventilated emergency department patients receiving post-intubation sedation after an educational initiative aimed at improving sedation practices in the ED
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Education — Nurses and physicians will be engaged regarding the clinical outcome data on the importance of ED-based sedation, and the objectives of the research. Education will include in-services and lectures focused on the importance of sedation protocols on patient outcome. The use of sedation will be evaluated throughout the study in order to better understand providers' perception of and experience with ED-based sedation protocols.
  Arms: After group
Other: Standard post intubation sedation practices — Usual care sedation provide in the ED
  Arms: Before group

SUMMARY:
The ED-SED Pilot is a multicenter, prospective, before-and-after study conducted on 344 mechanically ventilated emergency department patients at three academic medical centers: Washington University in St. Louis School of Medicine (St. Louis, MO), Cooper Hospital of Rowan University (Camden, NJ), and University of Iowa Carver College of Medicine (Iowa City, IA). The overall goal is to assess the feasibility of implementing targeted sedation (in terms of sedation depth) for mechanically ventilated ED patients in order to reduce the incidence of unnecessary deep sedation and improve clinical outcomes.

DETAILED DESCRIPTION:
The ED-SED Pilot is a multicenter, prospective, before-and-after study conducted on 344 mechanically ventilated ED patients at three academic medical centers. Patients in the before phase of the study will receive usual care after the initiation of mechanical ventilation. After 172 patients have been enrolled in the before phase, the investigators will begin educational initiatives to implement ED-based sedation protocols and order sets. The research team will educate providers on the importance of sedation protocols on patient outcome so that the existing protocols begin to be used effectively in the ED. This educational initiative will allow targeted sedation to be effectively used in the ED as well, allowing the intervention to be tested under real-world conditions. Participants in the after phase will also receive standard post-intubation care at the discretion of the treating team, though it will be after the educational initiative aimed at improving post-intubation sedation.

In order to more effectively use sedation in the ED, the investigators will collect voluntary and anonymous surveys from ED nurses and physicians to assess the potential facilitators and barriers to adherence to guideline-recommended sedation.

ELIGIBILITY:
Inclusion Criteria:

1. Mechanical ventilation via an endotracheal tube.
2. Age ≥ 18 years.

Exclusion Criteria:

1. Acute neurologic injury (stroke, intracranial hemorrhage, traumatic brain injury, cardiac arrest, status epilepticus, fulminant hepatic failure).
2. Ongoing neuromuscular blockade.
3. Death or transition to comfort measures within 24 hours.
4. Transfer to another hospital from the ED.
5. Chronic/home mechanical ventilation.
6. Transfer directly from the ED to the operating room.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1771 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2022-05-28 (Actual); Study Completion 2022-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Fuller, MD, Principal Investigator — Washington University School of Medicine
Locations (3):
- United States (3):
  - University of Iowa, Iowa City, Iowa
  - Washington University School of Medicine/Barnes-Jewish Hospital, St Louis, Missouri
  - Cooper University Hospital/Cooper Medical School of Rowan University, Camden, New Jersey

IPD SHARING:
Plan to Share IPD: No
Sharing of data generated by this trial is an important part of the proposed activities. Data will be shared with other investigators through academically established means, as necessary and appropriate. Datasets generated from the trial will be available from the overall study principal investigator on reasonable request. Collaboration with others investigators is encouraged. The results will be disseminated via publication in a peer-reviewed journal and presentation at national meetings.

REFERENCES:
- [Derived] Fuller BM, Pappal RD, Mohr NM, Roberts BW, Faine B, Yeary J, Sewatsky T, Johnson NJ, Driver BE, Ablordeppey E, Drewry AM, Wessman BT, Yan Y, Kollef MH, Carpenter CR, Avidan MS. Awareness With Paralysis Among Critically Ill Emergency Department Patients: A Prospective Cohort Study. Crit Care Med. 2022 Oct 1;50(10):1449-1460. doi: 10.1097/CCM.0000000000005626. Epub 2022 Jul 21. PMID 35866657
- [Derived] Fuller BM, Roberts BW, Mohr NM, Pappal RD, Stephens RJ, Yan Y, Carpenter C, Kollef MH, Avidan MS. A study protocol for a multicentre, prospective, before-and-after trial evaluating the feasibility of implementing targeted SEDation after initiation of mechanical ventilation in the emergency department (The ED-SED Pilot Trial). BMJ Open. 2020 Dec 16;10(12):e041987. doi: 10.1136/bmjopen-2020-041987. PMID 33328261

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Before Group | After Group
Started | 876 | 895
Completed | 196 | 219
Not Completed | 680 | 676

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Before Group | After Group | Total
Number analyzed (Participants) | 196 | 219 | 415
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 1 | 3
  Between 18 and 65 years | 120 | 134 | 254
  >=65 years | 74 | 84 | 158
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (18.4) | 57.4 (18.3) | 57.6 (18.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 90 | 161
  Male | 125 | 129 | 254
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 101 | 102 | 203
  Race: Black | 71 | 94 | 165
  Race: Hispanic | 14 | 18 | 32
  Race: Asian | 6 | 4 | 10
  Race: Other | 4 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 196 | 219 | 415

OUTCOME MEASURES:

1. Primary Outcome: Participant Recruitment
Description: Count of eligible participants included in study
Time Frame: Through study completion, an average of 1 year
Population: These numbers reflect the number of eligible participants who were included in the study for analysis (i.e. the final study population). As mentioned above in "Participant Flow", there were 1771 participants assessed for eligibility and 1356 were not eligible for the study. Therefore, the overall number of participants analyzed (i.e. 415) relects this.
Measure: Count of Participants; unit: Participants
Arm/Group | Before Group | After Group
Number analyzed (Participants) | 196 | 219
Participants | 196 | 219

2. Primary Outcome: Percentage of Patients With Richmond Agitation-Sedation Scale (RASS) Scores in Deep Sedation Range
Description: Deep sedation defined as RASS of -3 to -5
  Measure of Sedation via RASS. Scale: +4 Combative, +3 Very agitated, +2 Agitated, +1 Restless, 0 Alert and Calm, -1 Drowsy, -2 Light sedation, -3 Moderate sedation, -4 Deep sedation, -5 Unarousable
Time Frame: Up to 12 hours (during mechanical ventilation in the emergency department)
Measure: Count of Participants; unit: Participants
Arm/Group | Before Group | After Group
Number analyzed (Participants) | 196 | 219
Participants | 118 | 85

3. Primary Outcome: Reliability of Richmond Agitation-Sedation Scale (RASS) Measurements During Routine Care in the ED
Description: Interrater correlation coeficient. These were paired observations between study team members and ED nurses. It reflects the degree of agreement between independent observers.
Time Frame: Up to 12 hours (during mechanical ventilation in the emergency department)
Population: Reliability of RASS assessments was only assessed in the after group as an assurance that the protocol was being effectively implemented and RASS measured appropriately
Measure: Number (95% Confidence Interval); unit: ICC
Arm/Group | Before Group | After Group
Number analyzed (Participants) | 0 | 66
ICC |  | 0.88 [0.82 to 0.93]

4. Primary Outcome: Number of Participants With Adverse Events
Description: Inadvertent extubation, inadvertent device removal (e.g. central venous catheter, urinary catheter), awareness with paralysis events
Time Frame: Up to 12 hours (during mechanical ventilation in the emergency department)
Measure: Count of Participants; unit: Participants
Arm/Group | Before Group | After Group
Number analyzed (Participants) | 196 | 219
Participants | 8 | 11

5. Secondary Outcome: Ventilator-free Days
Description: To define, ventilator-free days equal: 1) 0 if patient dies within 28 days of mechanical ventilation; 2) 28 - x if successfully liberated from mechanical ventilation 'x' days after intubation; or 3) 0 if mechanical ventilation duration exceeds 28 days.
Time Frame: Up to 28 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Before Group | After Group
Number analyzed (Participants) | 196 | 219
days | 19.9 (10.6) | 22.0 (9.0)

6. Secondary Outcome: ICU-free Days
Description: To define, ICU-free days equal: 1) 0 if patient dies within 28 days of ICU admission; 2) 28 - x if successfully discharged from the ICU 'x' days after admission to the ICU; or 3) 0 if ICU length of stay exceeds 28 days.
Time Frame: Up to 28 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Before Group | After Group
Number analyzed (Participants) | 196 | 219
days | 18.1 (10.4) | 20.8 (8.7)

7. Secondary Outcome: Hospital-free Days
Description: To define, hospital-free days equal: 1) 0 if patient dies within 28 days of hospital admission; 2) 28 - x if successfully discharged from the hospital 'x' days after admission to the hospital; or 3) 0 if hospital length of stay exceeds 28 days.
Time Frame: Up to 28 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Before Group | After Group
Number analyzed (Participants) | 196 | 219
days | 14.3 (10.1) | 15.2 (9.2)

8. Secondary Outcome: Number of Participants With Delirium
Description: Delirium defined as being CAM-ICU positive as documented by bedside nurse during routine care.
Time Frame: Up to 7 days
Population: We recognize that the Overall Number of Participants Analyzed is not consistent with numbers provided in any of the rows in the Participant Flow module. The numbers analyzed for delirium reflect the fact that some patients either died or were discharged and therefore not eligible to be assessed for delirium during the time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Before Group | After Group
Number analyzed (Participants) | 167 | 198
Participants | 63 | 62

9. Secondary Outcome: Mortality
Description: Hospital mortality
Time Frame: Up to 28 days, or for the duration of hospitalization
Measure: Count of Participants; unit: Participants
Arm/Group | Before Group | After Group
Number analyzed (Participants) | 196 | 219
Participants | 40 | 22

ADVERSE EVENTS:
Time Frame: Serious adverse events related to care in the emergency department were collected up to 12 hours (during mechanical ventilation in the emergency department). These were reported as outcomes and include: inadvertent extubation, device removal, and awareness with paralysis. All-cause mortality was collected up to 28 days, or for the duration of hospitalization. Other (Not Including Serious) Adverse Events were collected up to 28 days, or for the duration of the hospitalization.
Description: Serious adverse events related to care in the emergency department were collected up to 12 hours (during mechanical ventilation in the emergency department). These were reported as outcomes and include inadvertent extubation, device removal, and awareness with paralysis.
  All-cause mortality was collected up to 28 days, or for the duration of hospitalization.
  Adverse Events were monitored/assessed without regard to the specific Adverse Event Term.
Arm/Group | Before Group | After Group
All-Cause Mortality (participants affected / at risk) | 40/196 | 22/219
Serious Adverse Events (participants affected / at risk) | 8/196 | 11/219
Other Adverse Events (participants affected / at risk) | 0/196 | 0/219
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Before Group (N=196) | After Group (N=219)
Inadvertent extubation, device removal, awareness with paralysis (Surgical and medical procedures) | 8 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-03): https://cdn.clinicaltrials.gov/large-docs/83/NCT04410783/Prot_SAP_000.pdf